CLINICAL TRIAL: NCT04524325
Title: Mechanisms of Blood Pressure Dysfunction in Transmen Receiving Testosterone
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding never received.
Sponsor: Yale University (Other)
Collaborators: The John B. Pierce Laboratory (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000027735
Record Dates: First submitted 2020-08-17; First posted 2020-08-24 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Transgender Men; Blood Pressure; Hyperandrogenism
Keywords: transgender; baroreflex; testosterone
MeSH Terms: conditions — Hyperandrogenism

STUDY DESIGN:
Intervention Model Description: There is 1 group of trans men (n=20) and 1 group of cisgender women (n=20). Study procedures, protocols, and measurements will be the same for both groups and performed and/or taken in a similar time period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trans men (Active Comparator): transgender men taking physiologic doses of testosterone for gender affirming hormone therapy
  Interventions: Other: Trans men
- control (No Intervention): cisgender women not receiving testosterone and with normal sex hormone levels

INTERVENTIONS:
Other: Trans men — We are studying the effects of testosterone taken by trans men on mechanisms of blood pressure control and comparing those results to cisgender women that have normal (ie lower) testosterone levels.
  Arms: Trans men

SUMMARY:
The purpose of this research is to explore the effects of chronic androgen exposure on sympathetic nervous system activity (SNSA) and baroreflex control of blood pressure responses in transgender men (trans men) taking gender affirming hormone therapy (HT). Blood pressure, baroreflex gain, and frequency of sympathetic responses to changes in blood pressure will be assessed in trans men and a control group of cisgender women. To fully understand HT effects on blood pressure regulation in trans men, it is crucial to understand how both SNSA, and the pattern of SNSA, can be influenced by high levels of androgen exposure in the female cardiovascular system, as well as how the two regulatory components may interact.

DETAILED DESCRIPTION:
The purpose of this research is to study how testosterone affects blood pressure control in trans men. High testosterone levels are detrimental to the female cardiovascular system in that higher levels are associated with increased blood pressure. Humans control blood pressure in the autonomic nervous system via the baroreflex mechanism. The arterial baroreflex is a key autonomic homeostatic mechanism involved in maintaining arterial blood pressure, and gain of the baroreflex is used as a measure of the sensitivity of sympathetic responses that act to restore acute blood pressure fluctuations. This autonomic regulation of blood pressure is also characterized by rhythmic activity (changes in cardiac frequency), which can be observed by recording sympathetic nerve traffic. When the female cardiovascular system is exposed to elevated androgens, baroreflex gain is impaired, and blood control is less efficient during an orthostatic challenge. However, to best understand the effect of a given stimulus on autonomic function, changes in frequency of the SNSA response must also be quantified in addition to the gain. Sympathetic control of arterial blood pressure is most effective in a narrow frequency range, and if this frequency range for responsiveness should narrow further, control of arterial blood pressure becomes less efficient and presents as dysfunction. The central hypothesis for this research is that dysregulation of blood pressure in trans men taking testosterone for gender affirming HT is a function of both reduced baroreflex gain and narrowed frequency-dependent relationship between arterial pressure and peripheral sympathetic vascular responsiveness. Specifically, these studies test the hypothesis that androgen supplementation with HT is associated with 1) lower baroreflex gain during a lower body negative pressure (LBNP) challenge, and 2) a narrowed response frequency range that precedes impaired sympathetic vascular response dynamics in trans men compared to control cisgender women.

Study procedures include an oral glucose tolerance test (OGTT), microneurography of the median nerve in the forearm to assess SNSA, and 2 LBNP challenges designed to examine baroreflex gain during static LBNP and then the frequency of SNSA during oscillating LBNP (OLBNP). Participants complete 3 visits for this study. Visit 1 is for informed consent procedures; Visit 2 is a pre-screening visit to complete the OGTT; Visit 3 is for experimental testing to assess gain and the frequency range. Blood pressure, heart rate and muscle SNSA (MSNA) are measured during LBNP and OLBNP. MSNA is recorded using 2 microelectrodes inserted through the skin of the forearm to record activity (firing) of the median nerve. Blood samples are taken via IV placement to measure insulin and glucose during the OGTT for Visit 2, and then sex hormones and catecholamines during Visit 3. Results from the group of young trans men will be compared to a control group of cisgender women matched for age and body mass index.

ELIGIBILITY:
Inclusion Criteria:

* Both groups (trans men and cisgender women) must be healthy and non-smoking. Control participants must be cisgender women with regular menses every 26-34 days. Trans men participants must be currently receiving testosterone for gender affirming hormone therapy where physiologic doses of exogenous Dihydrotestosterone have been administered (via injection or transdermal application) for at least 3 months as prescribed by their local endocrine provider as part of their clinically indicated hormone therapy. Doses can vary depending on the size and goals of each patient, but blood testosterone will be between 400-1000 ng/dl.

Exclusion Criteria:

* Subjects who smoke, have diabetes, or BP>140/90 will be excluded.
* Subjects will not be taking medications during the study, including any insulin-sensitizing or cardiovascular medications.
* Subjects are excluded if they have lost > 5 kg of weight within the past 6 months or perform high-intensity exercise > 3 times/week.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Transgender men will be recruited for participating in the experimental group; cisgender women will be recruited for participation in the control group.
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Muscle Sympathetic Nerve Activity (MSNA) | 3 hours
  MSNA is recorded continuously at rest and during O/LBNP protocols with a tungsten microelectrode (0.2 diameters insulated shaft tapered to an uninsulated tip of ~1-5 μm) inserted percutaneously into the median nerve. Multiunit, postganglionic MSNA is distinguished from other sources of nerve activity by the presence of spontaneous pulse synchronous bursts, increased activity when the subject holds their breath or clenches their first (stretches forearm muscles around median nerve), or if activity does not change when the skin is stimulated by light brushing or stroking (indicates lack of skin nerve activity). Bursts of MSNA at rest and during LBNP are quantified as total activity (AU/min), burst frequency (bursts/min) and burst incidence (bursts/100 heartbeats). The MSNA burst incidence is expressed in bursts/100 heartbeats to normalize for differences in heart rate among subjects.
Systolic Blood Pressure (SBP) | 3 hours
  SBP is measured continuously with a Finometer beat-to-beat blood pressure measurement system at rest and during O/LBNP protocols. Units are mm Hg.
Diastolic Blood Pressure (DBP) | 3 hours
  DBP is measured continuously with a Finometer beat-to-beat blood pressure measurement system at rest and during O/LBNP protocols. Units are mm Hg.
Mean Arterial Pressure (MAP) | 3 hours
  MAP at rest and during O/LBNP protocols is calculated as 1/3(SBP-DBP)+DBP using the beat-to-beat SBP and DBP measurements taken with the Finometer system. Units are mm Hg.
Sympathetic Baroreflex (BR) Gain | 3 hours
  Sympathetic BR gain is used as an index of sympathetic (neural) control of blood pressure, where gain is determined by the slope of the linear relationship between MSNA (burst/100 heartbeats) and DBP (mm Hg) at rest and during LBNP. The relationship produces a negative slope in that for a given subject, when DBP falls below the normal level sustained at rest, sympathetic activity increases to restore DBP back to that normal level. Thus, more MSNA bursts are observed at lower levels of DBP and vice versa. A steeper (more negative) slope suggests greater sensitivity of the baroreceptors to changes in blood pressure, and thereby more effective sympathetic control of blood pressure. A flatter slope suggests impaired BR sensitivity and blood pressure dysfunction, which is expected for the trans men group compared to cisgender women controls.
Frequency in the Neural Cardiovascular Control | 0.5 hours
  The frequency of SBP, DBP and heart rate during OLBNP is analyzed in Matlab in a linear time-invariant system (LTI) framework. Heart rate and BP measures taken during OLBNP are low-pass filtered (0.05 Hz estimated example) and corrected for end-effects using a Hamming window. The derived impulse responses (IRs) are 1/3rd octave smoothed before calculating the frequency power spectra (0.001-0.05 Hz estimated example). The power of DBP and SBP at the OLBNP frequency are anticipated to be independently inversely related to the efficiency of BP control. Further, the difference in heart rate and SBP, and in heart rate and DBP, power at those frequencies reflects the degree of autonomic function, analogous to baroreflex gain.
Electrocardiogram (ECG) | 3 hours
  A 3-lead ECG is continuously recorded at rest and during the O/LBNP protocols. The R-wave of the QRS complex of the ECG recording will be used for measures of pulse interval by determining the amount of time in seconds between the R-waves of 2 consecutive QRS complexes.

SECONDARY OUTCOMES:
Brachial Artery Mean Blood Flow Velocity | 3 hours
  Mean blood flow velocity in the brachial artery will be examined at rest and during LBNP using Doppler ultrasound velocimetry. Blood flow velocity spectra and arterial diameter are measured simultaneously with a Doppler probe and SonoScape S2 ultrasound system. The brachial artery is imaged with a 6.0-MHz linear array probe positioned at a 45° angle over the skin at the distal one-third of the upper arm. Brachial blood flow is expected to decrease as the level of LBNP increases and induces a greater orthostatic challenge. For example, blood flow would be highest at the -10LBNP stage and continually decrease during the following stages of -20, -30 and finally -40LBNP, where blood flow would be the lowest.
Cardiovagal Baroreflex (BR) Gain | 3 hours
  Cardiovagal BR gain is determined by the slope of the linear relationship between R-R Interval (seconds) and SBP (mm Hg) at rest and during LBNP. R-R Intervals are obtained from the ECG recording and SBP is obtained from the beat-to-beat measures taken by the Finometer.

IPD SHARING:
Plan to Share IPD: Undecided